CLINICAL TRIAL: NCT00280189
Title: A Prospective Study of Outcomes of Radiofrequency Ablation of Lung Tumors
Brief Title: Study of Outcomes of Radiofrequency Ablation of Lung Tumors
Status: Suspended | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: RITA Medical Systems (Industry)
Responsible Party: Principal Investigator, James Luketich, Professor, University of Pittsburgh
Other Study IDs: STUDY20050042; #02-033 (Other: UPCI)
Record Dates: First submitted 2006-01-18; First posted 2006-01-20 (Estimated); Last update posted 2025-04-16 (Actual); Status verified 2025-02

CONDITIONS: NSCLC; Pulmonary Metastases
Keywords: Radiofrequency ablation; Pulmonary malignancies; Primary lung cancer; Pulmonary metastasis; Primary lung tumors; Secondary lung tumors; Coagulation necrosis of soft tissue tumors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Radiofrequency ablation of pulmonary malignancies — Radiofrequency ablation is an inpatient procedure typically requiring one overnight stay in the hospital.
Behavioral: Quality of life assessment — Quality of life assessment is administered prior to the Radiofrequency ablation procedure and every 3 months for 1 year following the procedure.
Behavioral: Assessment of pain — Pain scores are obtained prior to the procedure, daily X 7 starting on the day of surgery, and then every 3 months for 1 year.

SUMMARY:
The purpose of this study is to assess short and long term outcomes after radiofrequency ablation (RFA) of pulmonary malignancies in patients who are not candidates for surgical resection. This study will evaluate the efficacy of RFA for the treatment of lung tumors by assessing its impact on local tumor control, progression free survival, overall survival, dyspnea score and quality of life (QOL).

DETAILED DESCRIPTION:
The use of RF ablation in pulmonary tissue is not new. However previous reports have primarily been descriptions of technique and early procedural outcomes. Follow-up studies have been lacking. This study will provide information on outcomes such as rates of clinical response, overall survival, progression-free survival, dyspnea and QOL.

The determination of the efficacy of this technique with this study could make an important contribution to the management of patients with pulmonary malignancies with high operative risk for resection. A minimally invasive alternative for tumor destruction could potentially improve quality of life by controlling local tumor progression and could provide longer survival when compared to current non-surgical options. This pilot study will determine the potential utility and effectiveness of RFA treatment of lung tumors, and whether to further evaluate this therapy in prospective randomized clinical trials compared to other conventional modalities.

Lung cancer is currently the most common cause of cancer-related death in the USA and represents the second most common malignancy in both men and women with 171,400 new cases in the year 1999. Unfortunately, the majority of patients present with advanced disease. Despite advances in the management of this disease, the best 5-year survival for stage I remains around 70% for patients who have undergone surgical resection. Complete resection provides the best chance for cure and remains the gold standard of therapy for patients with acceptable surgical risk.

The role of surgical resection of pulmonary metastasis in selected patients is widely accepted, and a survival advantage of aggressive surgical therapy has been demonstrated. Surgical series have demonstrated 5-year survival of 25-42% in the surgical treatment of pulmonary metastasis from different primaries including colorectal cancer osteogenic sarcoma, melanoma, and others. In a prospective study of 5,206 cases of lung metastasectomy, the International Registry of Lung Metastases reported an actuarial survival of 36% at 5 years and 26% at 10 years. These results compared favorably with those who had an incomplete resection achieving a survival of 13% at 5 years and 7% at 10 years.

The standard resections for primary lung cancer include lobectomy or pneumonectomy depending on the size and location of the tumor. Limited resections, including segmentectomy or wedge resection of the lung, are the standard treatment for limited metastases and are good alternatives for patients with primary lung cancer and poor lung function who cannot tolerate a larger resection. However, a prospective randomized trial to address the role of limited resection for primary lung cancer was performed by the Lung Cancer Study Group in 276 patients with T1N0 NSCLC. Patients in the limited resection group suffered a 50-75% increase in local recurrence rate, but no survival difference was seen between the two groups. Limited resection however should continue to be viewed as a good option for metastasectomy but a compromising operation for primary lung cancer.

The treatment options for patients with pulmonary malignancies who have severe comorbidities or poor pulmonary function are limited. These patients are many times not considered for surgical resection because of the excessive risk of undergoing an invasive operation and are often treated with external beam radiation and/or chemotherapy. In the case of pulmonary metastases occurring after previous pulmonary resection, further resection is sometimes not feasible due to limited residual pulmonary parenchyma or dense adhesions.

After the widespread application of radiofrequency ablation (RFA) for the destruction of unresectable liver tumors, this technique has been considered as an alternative therapy for the ablation of other solid tumors. The initial experience in the treatment of lung tumors with RFA indicates that the technique appears to be safe and feasible for ablation of peripheral lung nodules.

The U.S. Food and Drug Administration approved RFA for coagulation necrosis of soft tissue tumors. In addition, RFA has been widely used for treatment of pulmonary nodules in France, Germany, Japan, Korea, and the People's Republic of China.

Radiofrequency ablation systems are comprised of three components: a radiofrequency generator, an active electrode, and dispersive electrodes. The RF energy is introduced into the tissue via the active electrode. As the RF energy (alternating current) moves from the active electrode to the dispersive electrode (i.e., the electrosurgical return pad) and then back to the active electrode, the ions within the tissue oscillate in an attempt to follow the change in the direction of the alternating current. This movement results in frictional heating of the tissue, and as the temperature within the tissue becomes elevated beyond 60°C, cells begin to die. It is this phenomenon that causes the region of necrosis surrounding the electrode.

The advantage of such a thermal intervention system is the capacity to heat tissue to a lethal temperature in a specific anatomic location. The advantages of such a procedure in the treatment of non-resectable hepatic and renal lesions are reduced surgical trauma, shorter procedure time, shorter hospitalization, and a faster recovery time. In the treatment of lung nodules, this allows for destruction of lung tumors with minimal damage to surrounding normal lung tissue.

Coagulation necrosis of soft tissue due to RF ablation has been reported in liver, kidney, breast, and lung tissues. Radiofrequency ablation of primary and metastatic hepatic lesions has been reported to result in necrosis encompassing 70% to 98% of tumors treated. To date, little has been reported on the use of RF ablation to address pulmonary nodules. In a presentation of three case studies, follow-up CT imaging noted that cells within the region of the thermal lesions were fibrotic and in only one of the three patients was residual disease detected. Using positron emission tomography (PET) imaging of the lung, a series of ten patients noted that within the boundaries of the thermal lesions there was no evidence of metabolic activity.

A pre-clinical study was undertaken in a porcine model in order to determine the capacity of RF energy to induce necrosis of lung tissue. Using differing power settings and length of application times, it was determined that the thermal lesions produced in the porcine lung tissue were complete and entire, with no procedure-related complications. Animals survived to 3, 7 and 28 days post-RF ablation were active and showed no evidence of detrimental effects of the RF-induced necrosis on respiratory capacity or function. The regions of necrosis were affected by conductive heat loss via air and blood flow and the presence of bronchi, which resulted in invagination of the thermal lesion boundary; however, all cells within the boundaries were nonviable.

Determining the effectiveness of the RF ablation usually involves follow-up computed tomography (CT) scans. CT imaging provides an assessment of tissue changes following an ablation, which can manifest as central cavitation of the lesion with decreased tissue density measured by a decrease in Hounsfield units (Hu). As complementary modality, positron emission tomography (PET) can be used to determine tissue viability within the lesion, which can be useful in the follow-up of these patients. In particular, patients with questionable response to RFA as determined by CT scan can benefit from PET scanning, by determining the presence of residual disease. The patient is injected with a radio-labeled sugar (typically 18 Fluoro-deoxyglucose or FDG) prior to the PET scan and viability is determined based upon the uptake of the FDG by cells, since FDG is taken up by cells with high metabolic activity, such as tumors, infection, or inflammation. In a small pilot study, monitoring with PET noted no viable tissue within the boundaries of the thermal lesions induced in pulmonary nodules.

In the investigators' initial experience at the University of Pittsburgh Medical Center, they treated 18 patients with RFA and included primary and metastatic lung tumors. Selected patients were not candidates for complete surgical resection based on surgical risk, multiple lesions, poor pulmonary reserve or refusal of further surgery. Twenty-eight lung nodules were treated with RFA in 18 patients (12 male, 6 female). Tumors included metastatic carcinoma (9), sarcoma (6) or lung cancer (3). Mean age was 52 years (range, 27-95). Thoracic surgeons performed RFA by mini-thoracotomy (5) or CT-guided percutaneously (13) under general anesthesia in the operating room. In both approaches, the patient was positioned in the lateral decubitus position. In the CT-guided procedures we employ the services of a CT technician and the thoracic surgeon places a small finder needle into the center of the lung nodule. The surgeon confirms successful central placement of the finder needle during CT imaging, and the LeVeen™ needle electrode size is chosen according to the diameter of the target lesion. The needle electrode has a diameter of 14 gauge with a 15 cm shaft length and is introduced in the center of the lesion under CT guidance. Several applications in different locations within the lesion may be required for larger masses, with the therapy beginning at the most distal area and progressing proximally. Chest tubes were required in 46% (n=13) of percutaneous procedures. Mean length of stay was 3 days (range, 1-7 days). Complications included recurrent pneumothorax (1/18), pneumonitis (6/18), small pleural effusion (7/18) and transient renal failure (1/18). One death occurred from hemoptysis 19 days post-RFA of a central nodule. This patient had also received recent brachytherapy. After a mean follow-up of 4 months (range, 1-11 months), computed tomography revealed resolution with decreased density of treated sites less than 4 cm. Six patients (33%) died of progressive metastatic disease during the follow-up period.

Even though RFA has been used to treat lung tumors in over 300 patients worldwide, there is still a need to further define the role of RFA for pulmonary malignancies. In particular the effects of RFA on dyspnea and quality of life as well as follow-up studies are lacking.

ELIGIBILITY:
Inclusion Criteria:

* Have stage I or II primary lung cancer and who are felt not to be candidates for resection based upon co-morbid disease or who refuse lung resection.
* Have metastatic tumors to the lung, and who meet criteria for metastasectomy but who are felt not to be candidates for resection of all metastases. All metastases should be treatable by RFA alone or in combination with resection.
* Have positive tissue diagnosis by previous resection (less than 6 months) or by radiologic biopsy.
* Have clinically suspicious disease defined as a new lesion on chest CT or a suspicious PET scan.
* Have RF ablation target lesions of 4 centimeters or less in diameter.

Exclusion Criteria:

* If the lesion is centrally located, less than 3 centimeters from the hilum.
* If the target lesion is greater than 4 centimeters in diameter.
* If the lesion is metastatic and the primary site is not controlled.
* If extra-thoracic metastatic disease is present.
* If there are more than 3 tumors in one lung.
* If there are greater than 6 metastatic tumors in total (bilateral).
* If it is felt that all metastases cannot be treated by RFA alone or in combination with resection.
* If the patient is pregnant or nursing at the time of the procedure.
* If the patient has malignant pleural effusion.
* If the patient is unwilling or unable to provide consent for the procedure.
* If the patient is less than 18 years of age (the short form [SF]-36 is not designed for patients less than 18 years of age).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seeking minimally invasive treatment for pulmonary malignancies.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2003-09; Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Assess overall survival, progression-free survival and clinical response after RFA | Until disease progression or death

SECONDARY OUTCOMES:
To characterize QOL before and after RFA treatment | Every 3 months for 1 year then annually
To assess procedure related outcomes after RFA of lung tumors, in particular, measuring length of stay, morbidity and mortality and requirements for chest tube drainage | Within 30 days of RFA procedure

CONTACTS AND LOCATIONS:
Overall Officials: James Luketich, MD, Principal Investigator — UPMC - Department of Cardiothoracic Surgery
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided